CLINICAL TRIAL: NCT01767233
Title: Prophylactic Pancreatic Duct Stenting in Acute Necrotizing Pancreatitis: a Prospective Randomized Controlled Multicenter Study
Brief Title: Prophylactic Pancreatic Duct Stenting in Acute Necrotizing Pancreatitis
Acronym: ERPNEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36/2010
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Acute Necrotizing Pancreatitis
Keywords: Acute necrotizing pancreatitis; ERCP; Pancreatic stenting
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pancreatic stenting (Experimental): Pancreatic stenting versus observation
  Interventions: Procedure: ERCP and pancreatic stenting

INTERVENTIONS:
Procedure: ERCP and pancreatic stenting

SUMMARY:
Since the majority of patients with necrotizing pancreatitis will experience a leak from the pancreatic duct during their course of disease resulting in intra- and peripancreatic fluid collections, it is reasonable to hypothesize that placement of a ductal stent may prevent some of the late complications and morbidity associated with pancreatic necrosis. This prospective, randomized, controlled multicenter trial investigates the role of early prophylactic ductal stenting in acute necrotizing pancreatitis.

The purpose of the study is to determinate the safety and feasibility of early prophylactic pancreatic duct stenting in necrotizing pancreatitis in reducing complications, length of stay in hospital and in in-tensive care unit compared to the traditional treatment.

ELIGIBILITY:
Inclusion Criteria:

In patients with suspected necrotizing pancreatitis a pancreatic protocol 3-phase contrast enhanced (CE) CT shall be performed. Since a very early CT may underestimate the extent of pancreatic necro-sis, it is recommended to wait at least 72 hours after the onset of symptoms before CT is done. The CECT may be repeated if the initial CT shows no necroses and the clinical course continues to indicate a severe case.

MRI may be used instead of CT in case of contraindication to intravenous contrast due to renal failure.

If CECT reveals pancreatic necrosis affecting the head, neck, or body of pancreas and the necrosis is suspected to include the main pancreatic duct an informed consent to participate in the study is ob-tained, after which the patient will be randomized to either a) the control group with traditional treat-ment (i.e. at the discretion of each participating center) or to b) the intervention group with same treatment as in the control group plus ERP and PD-stenting. Patients with isolated necrosis of the tail will not be included in the study.

Exclusion Criteria:

All consecutive patients (age between 18-75 years) admitted to the participating centers for acute pan-creatitis with an area of non-enhancing pancreatic parenchyma on CT believed to represent necrosis are prospectively enrolled in the study. At initial presentation the age, gender, etiology of the pancreatitis, clinical and laboratory findings will be recorded. Patients with malignancies and patients from whom an informed consent to participate in the study cannot be obtained will be excluded.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The need for percutaneous, endoscopic, laparoscopic, or open surgical drainage and/or debridement after randomization. | 12 months
  The indications for drainage/debridement are:
  1. Infection
  2. Gastro-intestinal or bile duct obstruction
  3. Pain caused by pancreatic or peripancreatic collection(s)
  4. Leakage of pancreatic juice (i.e. ascites or pleural fluid with an amylase content greater than 3 times the serum amylase activity)

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Oulu, Finland

REFERENCES:
- [Derived] Karjula H, Nordblad Schmidt P, Makela J, Liisanantti JH, Ohtonen P, Saarela A. Prophylactic pancreatic duct stenting in severe acute necrotizing pancreatitis: a prospective randomized study. Endoscopy. 2019 Nov;51(11):1027-1034. doi: 10.1055/a-0865-1960. Epub 2019 Mar 20. PMID 30895583